CLINICAL TRIAL: NCT00639730
Title: Use of the Atkins Diet for Children With Sturge Weber Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Vascular Birthmarks Foundation (Other)
Responsible Party: Eric Kossoff MD, Johns Hopkins School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00003359
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Epilepsy; Sturge Weber Syndrome
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy; Sturge-Weber Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): This is open-label - all patients are placed on the diet. There is no control or placebo arm.
  Interventions: Dietary Supplement: modified Atkins diet

INTERVENTIONS:
Dietary Supplement: modified Atkins diet — High fat, low carbohydrate diet

SUMMARY:
This research is being done to find out if the Atkins Diet can be used safely and effectively to reduce seizures in children who have Sturge Weber syndrome.

The ketogenic diet is a proven therapy for epilepsy, but can be difficult to use in children. The Atkins Diet is a high fat, high protein, low carbohydrate diet introduced in the 1970s to help with weight loss. It is different from the ketogenic diet in four major ways: no calorie restriction, no fluid restriction, no protein restriction, and is easy to start outside the hospital. People on the Atkins Diet become ketotic (produce high levels of ketones, a certain substance in the body), like patients on the ketogenic diet, and the investigators believe this may lead to seizure control.

Children aged 2-18 with Sturge Weber syndrome and seizures at least monthly, who have used at least two anti-seizure drugs may join. 5 children in total will be enrolled.

DETAILED DESCRIPTION:
If you agree to be in this study, we will ask you to do the following things:

Before the diet is started:

* We will ask you to keep track of your child's seizures daily for 2 weeks before starting the Atkins diet and provide us with a 3-day food record as well.
* Baseline blood (about 2 teaspoons) and urine work will be obtained.
* We will give you a free copy of a carbohydrate-counting guide.
* You will be asked to fill out a 3-day food record.

On the diet:

* Give your child a daily calcium supplement and multivitamin.
* Keep a daily seizure log.
* Check urine for ketones (to make sure the diet is working) and specific gravity (to make sure your child is well hydrated) twice a week and when you come to clinic.
* We will ask you to weigh your child at home every week, and we will weigh him or her when you come into clinic too.
* Do not fluid restrict your child; please give plenty of carbohydrate-free fluids.
* You will give 20 grams per day of carbohydrates. We will give you instructions on how to measure daily intake of carbohydrates.
* We will not change medications for the first three months. Do not change your child's seizure medicines without checking with our doctors.
* For the first three months, we ask you to avoid store-bought low-carbohydrate products (as they can have more carbohydrates than advertised).

After being on the diet for one month, Dr. Kossoff will contact you by telephone to discuss how your child is doing. You can also speak with one of our dietitians. We will discuss the 3-day food record with you

You will be asked to come to the clinic (outpatient center, 5th floor) for two follow-up visits:

1. after being on the diet for 3 months and
2. after being on the diet for 6 months.

During these visits you will meet with one of our doctors and a dietitian. We will review your child's seizure control and health. We may obtain blood (about 2 teaspoons). We will check your child's urine for ketones and specific gravity.

If the diet is helping beyond 6 months, we will help your child continue on the diet with clinic visits and labs as necessary, at a carbohydrate amount that is most helpful.

ELIGIBILITY:
Inclusion Criteria:

* 2-18 years
* Sturge Weber syndrome
* Monthly seizures (at least)
* Tried at least two anticonvulsants

Exclusion Criteria:

* Prior use of the Atkins or ketogenic diets
* Patients with non-epileptic seizures (pseudoseizures) will be excluded
* Patients that are pregnant or become pregnant during the study will be excluded
* High cholesterol

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2006-05; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Seizures | 6 months
  Seizure frequency will be compared to baseline (pre-Diet).

SECONDARY OUTCOMES:
Ketosis | 6 months
Safety (stroke like events) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric H Kossoff, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kossoff EH, Turner Z, Bluml RM, Pyzik PL, Vining EP. A randomized, crossover comparison of daily carbohydrate limits using the modified Atkins diet. Epilepsy Behav. 2007 May;10(3):432-6. doi: 10.1016/j.yebeh.2007.01.012. Epub 2007 Feb 26. PMID 17324628
- [Background] Kossoff EH, McGrogan JR, Bluml RM, Pillas DJ, Rubenstein JE, Vining EP. A modified Atkins diet is effective for the treatment of intractable pediatric epilepsy. Epilepsia. 2006 Feb;47(2):421-4. doi: 10.1111/j.1528-1167.2006.00438.x. PMID 16499770